CLINICAL TRIAL: NCT04817761
Title: SPARK-ALL: A Multi-center, Open-label, Single-arm Phase 2/3 Trial Evaluating the Safety and Pharmacokinetics of Calaspargase Pegol for Treatment of Adults Aged 22 To >65 Years With Newly-diagnosed Philadelphia-negative ALL.
Brief Title: SPARK-ALL: Calaspargase Pegol in Adults With ALL
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Institut de Recherches Internationales Servier (Other)
Collaborators: ADIR, a Servier Group company (Industry)
Responsible Party: Sponsor
Organization: Servier (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL2-95015-001
Record Dates: First submitted 2021-03-15; First posted 2021-03-26 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: Acute Lymphoblastic Leukemia; ALL; Ph-negative B-cell and T cell ALL; Philadelphia-negative ALL; Calaspargase Pegol; Asparlas; Adult; Acute Lymphocytic Leukemia; Newly diagnosed ALL; Untreated ALL
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma | interventions — calaspargase pegol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Calaspargase pegol (S95015) (Experimental)
  Interventions: Drug: Calaspargase pegol (S95015)

INTERVENTIONS:
Drug: Calaspargase pegol (S95015) — Part 1: S95015 will be administered at dose of 2000 U/m2, 1500 U/m2 or 1000 U/m2 (dose level based on age and BMI) via a 2-hour intravenous infusion at Day 4 (or 5, or 6) of the induction phase, Days 15 and 43 of the consolidation phase, Day 22 of the interim maintenance phase and Days 4 (or 5, or 6) and 43 of the delayed intensification phase. S95015 starting doses for age and BMI groups will be confirmed.
  Patients will receive premedication prior to calaspargase pegol administration (acetaminophen, histamine-1 blocker, and corticosteroids to prevent hypersensitivity reaction) and other backbone chemotherapy agents based on the CALGB 10403 protocol treatment regimen.
  Part 2: Patients aged 22 to 39 years + BMI ≤ 35 kg/m2 will be treated with S95015 1750 U/m2.
  Patients aged 40 to < 55 years + BMI ≤ 35 kg/m2 will be treated with S95015 1500 U/m2, unchanged from Part 1. Patients 55 years or older or those with a BMI greater than 35 kg/m2 will no longer be enrolled into Part 2.

SUMMARY:
The purpose of this phase 2/3 study is to confirm the recommended doses and to evaluate the safety and pharmacodynamics of Calaspargase pegol for the treatment of adult patients with Philadelphia-negative Acute Lymphoblastic Leukemia.

DETAILED DESCRIPTION:
The study will be conducted in 2 parts. Part 1 is a dose confirmation run-in period. Part 2 will enroll the remaining participants at the dose as confirmed or recommended in Part 1.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥22 and <55 years with newly-diagnosed and cytologically confirmed and documented Philadelphia-negative B-cell or T-cell ALL by World Health Organization (WHO) classification (2016).
* Eastern Cooperative Oncology Group performance status (ECOG PS) 0 to 2.
* No prior therapy for ALL such as chemotherapy and radiation therapy before signing the informed consent except for limited treatment (≤7 days) with corticosteroids or hydroxyurea and a single dose of intrathecal cytarabine.

Exclusion Criteria:

* Patients with Philadelphia chromosome positive ALL, Burkitt's leukemia, mixed lineage/mixed phenotype acute leukemia, and acute undifferentiated leukemia per WHO classification (2016).
* Patients with Down syndrome.
* Patients with Hepatitis B (positive for HBs antigen), and Hepatitis C (HCV antibody) at inclusion
* Participants known to be HIV-positive.
* Known history of non-gallstone-related pancreatitis.
* Known severe hepatic impairment (bilirubin >3 x upper limit of normal [ULN]; transaminases >10 times ULN.
* Pre-existing history of hepatic veno-occlusive disease (VOD).
* Age ≥ 55 years.
* BMI > 35 kg/m2.

Ages: 22 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 122 (Estimated)
Dates: Start 2021-07-07 (Actual); Primary Completion 2025-03-21 (Actual); Study Completion 2026-02-09 (Estimated)

PRIMARY OUTCOMES:
Adverse Events (AEs) (Part 1) | From signing the ICF through 30 days after the Calaspargase pegol administration at Day 4 (or Day 5 or Day 6) in the Remission Induction phase.
  Including Treatment-emergent adverse events (TEAEs), adverse events of special interests (AESI); laboratory tests; vital signs; serious adverse events (SAEs) and AE. AEs recoded and evaluated throughout the study in accordance with NCI CTCAE criteria 5.0.
Adverse Events (AEs) (Part 2) | From signing the ICF through 30 days after the last dose of the study drug in Delayed Intensification phase.
  Including Treatment-emergent adverse events (TEAEs), adverse events of special interest (AESI); laboratory tests; vital signs; serious adverse events (SAEs) and AEs. AEs recoded and evaluated throughout the study in accordance with NCI CTCAE criteria 5.0.
Plasma Asparaginase Activity (PAA) level (Part 1) | Days 4, 5, 6 (Remission Induction phase) for PAA samples. Days 11, 18, 25 (Remission Induction phase) for TDM samples.
  Assessment of PAA in Part 1 is based on population modeling analysis.
Nadir Plasma Asparaginase Activity (NPAA) (Part 2) | Day 64 (Remission Consolidation Phase).
  NPAA level ≥0.1 U/mL 21 days after the Remission Consolidation Phase Day 43 dose.

SECONDARY OUTCOMES:
Plasma Asparaginase Activity (PAA) level ≥0.1 U/mL at any time during Remission Induction phase and post- Remission Induction phase, respectively (Part 2) | Days 4-5-6 & 11-18-25 (Remission Induction); Days 15-16-43-44 & 22-29-36-50-57-64 (Consolidation); Days 22-23 & 29-36-43 (Interim Maintenance); Days 4-5,43-44 & 11-18-25-50-57-64 (Delayed Intensification) for PAA & TDM samples respectively.
  Pharmacodynamics criterion.
Plasma Asparaginase Activity (PAA) level ≥0.025, ≥0.1, ≥0.2, or ≥0.4 U/mL at predefined time points during Remission Induction phase and post- Remission Induction phase, respectively (Part 2) | Days 4-5-6 & 11-18-25 (Remission Induction); Days 15-16-43-44 & 22-29-36-50-57-64 (Consolidation); Days 22-23 & 29-36-43 (Interim Maintenance); Days 4-5-43-44 & 11-18-25-50-57-64 (Delayed Intensification) for PAA & TDM samples respectively.
  Pharmacodynamics criterion.
PAA-derived maximum concentration (Cmax) after the Remission Induction Phase Day 4 dose (Part 1 and 2). | Days 4, 5, 6 & 11, 18, 25 (Remission Induction); for PAA & TDM samples respectively.
  PAA-derived Cmax are based on population modeling analysis.
PAA-derived Area Under the PAA-Time Curve From Time 0 to Day 21 (AUC 0-21) after the Remission Induction Phase Day 4 dose (Part 1 and 2). | Days 4, 5, 6 & 11, 18, 25 (Remission Induction); for PAA & TDM samples respectively.
  PAA-derived AUC 0-21 are based on population modeling analysis.
Minimal residual disease (MRD) (Part 1 and 2) | End of remission induction phase (Day 29).
  Efficacy criterion.
Complete remission (CR) (Part 1 and 2) | Day 29 remission induction therapy
  Morphologic complete remission rate (CR), morphologic complete remission rate with incomplete blood count recovery (CRi).
Survival (Part 1 and 2) | Through study completion an average of 3 months.
  * 1-year EFS (event-free survival), DFS (disease-free survival) and OS (overall survival)
  * 2-year EFS, DFS, OS
  * 3-year EFS, DFS, OS.
Anti-drug (calaspargase pegol) antibody (ADA) development (Part 1 and 2) | D4, D18, D29 (Remission Induction Phase), D15, D43 (Remission Consolidation Phase), D22 (Interim Maintenance Phase), D4, D43 (Delayed Intensification Phase), Day 365 (±7) after the first dose, Day 30 after the last dose if discontinuation.
  Immunogenicity criterion.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J. DeAngelo, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute, Boston, MA
Locations (19):
- United States (19):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Univeristy of California, Los Angeles, California
  - University of California Irvine Health (UCI Health), Orange, California
  - University of Miami Health System - Sylvester Comprehensive Cancer Center, Miami, Florida
  - University of Chicago Medicine, Chicago, Illinois
  - University of Kansas Cancer Center - Richard and Annette Bloch Cancer Care Pavilion, Westwood, Kansas
  - University of Maryland Greenbaum Cancer Center, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Dana Farber Cancer Institute, Weymouth, Massachusetts
  - Northwell Health Cancer Institute, Lake Success, New York
  - NYU Langone/Laura and Isaac Perlmutter Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Health & Science University (OHSU), Portland, Oregon
  - Jefferson Health, Philadelphia, Pennsylvania
  - Baptist Clinical Research Institute, Memphis, Tennessee
  - Intermountain Healthcare (IHC), Salt Lake City, Utah
  - University of Washington/Seattle Cancer Care Alliance/Fred Hutch, Seattle, Washington
  - West Virginia University Cancer Institute, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: Yes
Qualified scientific and medical researchers can request access to anonymized patient-level and study-level clinical trial data.
  Access can be requested for all interventional clinical studies:
  * used for Marketing Authorization (MA) of medicines and new indications approved after 1 January 2014 in the European Economic Area (EEA) or the United States (US).
  * where Servier is the Marketing Authorization Holder (MAH). The date of the first MA of the new medicine (or the new indication) in one of the EEA Member States will be considered for this scope.
  In addition, access can be requested for all interventional clinical studies in patients:
  * sponsored by Servier
  * with a first patient enrolled as of 1 January 2004 onwards
  * for New Chemical Entity or New Biological Entity (new pharmaceutical form excluded) for which development has been terminated before any Marketing authorization (MA) approval.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After Marketing Authorisation in EEA or US if the study is used for the approval.
Access Criteria: Researchers should register on Servier Data Portal and fill in the research proposal form. This form in four parts should be fully documented. The Research Proposal Form will not be reviewed until all mandatory fields are completed.
URL: https://clinicaltrials.servier.com/

REFERENCES:
- [Background] Stock W, Park JH, Emadi A, Abdul-Hay M, Cassaday RD, Pullarkat VA, Webster J, Pandya SS, Mogul MJ, Shvenke Y, Zhu JJ, Tessier A, DeAngelo DJ. Safety and Pharmacokinetics of Calaspargase Pegol in Adults with Newly Diagnosed Philadelphia-Negative ALL: A Phase 2/3 Study. Blood. 2021 Nov 23;138(Supplement 1):4406. doi: https://doi.org/10.1182/blood-2021-149463
- [Derived] Aldoss I, Ali A, Cassaday RD, Curran EK, Luskin MR, Maese LD, Orgel E, Douer D. Optimizing Asparaginase Treatment for Adolescent and Young Adult (AYA) Patients With Acute Lymphoblastic Leukemia: US Consensus Panel Recommendations. Am J Hematol. 2026 Jan;101(1):41-55. doi: 10.1002/ajh.70103. Epub 2025 Oct 11. PMID 41074700
- See also: Find Results on Servier Clinical Trial Data website — https://clinicaltrials.servier.com/
- Available data/document: Individual Participant Data Set — https://clinicaltrials.servier.com/
- Available data/document: Study Protocol — https://clinicaltrials.servier.com/
- Available data/document: Statistical Analysis Plan — https://clinicaltrials.servier.com/
- Available data/document: Informed Consent Form — https://clinicaltrials.servier.com/
- Available data/document: Clinical Study Report — https://clinicaltrials.servier.com/
- Available data/document: Study-level clinical trial data — https://clinicaltrials.servier.com/